CLINICAL TRIAL: NCT06718361
Title: Assessing Environmental Oxygen Levels During Artificial Ventilation and Oxygen Therapy: Prospective Observational Study
Brief Title: Environmental Oxygen Levels During Artificial Ventilation and Oxygen Therapy
Status: Completed | Type: Observational
Sponsor: David Peran, PhD, FERC (Other)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Sponsor-Investigator, David Peran, PhD, FERC, Deputy director, Zdravotnicka Zachranna Sluzba Karlovarskeho Kraje, P.O.
Organization: Zdravotnicka Zachranna Sluzba Karlovarskeho Kraje, P.O. (Other)
Other Study IDs: ZZSKVK-01-2024
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Oxygen Delivery; Intubation; Airway Control; Concentration
Keywords: oxygen; concentration of oxygen; risk of fire; airway management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- O2 mask: Delivering oxygen via face mask with different oxygen flow (5, 10, 15 l/min).
  Interventions: Other: Oxygen levels measurement (%)
- Bag mask ventilation: Delivering oxygen via bag mask ventilation
  Interventions: Other: Oxygen levels measurement (%)
- Supraglotic airway: Delivering oxygen via laryngeal mask with bag or mechanical ventilation
  Interventions: Other: Oxygen levels measurement (%)
- Orotracheal intubation: Delivering oxygen via orotracheal tube with bag or mechanical ventilation
  Interventions: Other: Oxygen levels measurement (%)
- High-Flow Nasal Oxygenation: Oxygen delivery via high-flow nasal oxygenation
  Interventions: Other: Oxygen levels measurement (%)

INTERVENTIONS:
Other: Oxygen levels measurement (%) — Measuring levels of oxygen in the environment around the patient in %.

SUMMARY:
European Resuscitation Council 2021 Guidelines and Advanced Life Support Provider Courses teach that the oxygen supply must be removed from the patient during defibrillation to the distance of minimum of 1 meter. Scientific articles describe few incidents of fire during defibrillation in oxygen - enriched atmospheres.

The study aims to performed a series of measurement of the oxygen concentration in the environment around the patient with different airway management used and ventilation provided.

ELIGIBILITY:
Inclusion Criteria:

* patients at the intensive care unit bed or on the operating theatre with oxygen therapy prescribed/indicated

Exclusion Criteria:

* no oxygen therapy started
* situation not allowing measurement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients undergoing oxygen therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Oxygen levels | From the initiation of oxygen therapy at the start of anesthesia induction until the completion of oxygen therapy at the end of the procedure (ranging from 30 minutes to 6 hours), oxygen concentration will be assessed continuously.
  The oxygen levels in percentage

SECONDARY OUTCOMES:
Normal oxygen levels after the end of oxygen therapy | From the end of oxygen therapy at the completion of procedure until the reappearance of normal oxygen levels (21%), assessed continuously, up to 10 minutes.
  Time till the normal level of oxygen is reached after the end of oxygen therapy

CONTACTS AND LOCATIONS:
Overall Officials: David Peran, PhD, Principal Investigator — Zdravotnicka Zachranna Sluzba Karlovarskeho Kraje, P.O.
Locations (1):
- FNKV University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
All data will be part of the future publication.

REFERENCES:
- [Background] Robertshaw H, McAnulty G. Ambient oxygen concentrations during simulated cardiopulmonary resuscitation. Anaesthesia. 1998 Jul;53(7):634-7. doi: 10.1046/j.1365-2044.1998.410-az0512.x. PMID 9771170
- [Background] Theodorou AA, Gutierrez JA, Berg RA. Fire attributable to a defibrillation attempt in a neonate. Pediatrics. 2003 Sep;112(3 Pt 1):677-9. doi: 10.1542/peds.112.3.677. No abstract available. PMID 12949302
- [Background] Miller PH. Potential fire hazard in defibrillation. JAMA. 1972 Jul 10;221(2):192. No abstract available. PMID 5067634
- [Background] Cantello E, Davy TE, Koenig KL. The question of removing a ventilation bag before defibrillation. J Accid Emerg Med. 1998 Jul;15(4):286. doi: 10.1136/emj.15.4.286. No abstract available. PMID 9681318
- [Background] Barker SJ, Polson JS. Fire in the operating room: a case report and laboratory study. Anesth Analg. 2001 Oct;93(4):960-5. doi: 10.1097/00000539-200110000-00031. PMID 11574364
- [Background] Hummel RS 3rd, Ornato JP, Weinberg SM, Clarke AM. Spark-generating properties of electrode gels used during defibrillation. A potential fire hazard. JAMA. 1988 Nov 25;260(20):3021-4. PMID 3184368